CLINICAL TRIAL: NCT03853226
Title: Cardiac Afterload Indices Measured in Ascending and Descending Aorta: Rational for the Use of Velocity-Pressure Loop in the Operating Room
Brief Title: Rational for the Use of Velocity-Pressure Loop in the Operating Room
Acronym: VPLOOP
Status: Completed | Type: Observational
Sponsor: Joaquim MATEO (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Sponsor-Investigator, Joaquim MATEO, MD, Hopital Lariboisière
Organization: Hopital Lariboisière (Other)
Other Study IDs: SRLF 11-356
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Radiography; Interventional
Keywords: After-load cardiac performance; high cardiovascular risk; surgical patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: All monitoring — For all patients, data from trans-esophageal Doppler, trans-thoracic echocardiography (TTE) and hemodynamic data are collected at the end of the procedure. During catheter withdrawal, pressure waveforms are recorded at two predefined aortic locations: in the ascending aorta and in the descending thoracic aorta just in front of the esophageal Doppler probe.

SUMMARY:
In surgical patients considered with "high cardiovascular risk", by their field or by the nature of their intervention, it is recommended to use hemodynamic monitoring including a continuous measurement device of arterial pressure and cardiac output (CO). However, targeting mean arterial pressure (MAP) with boluses of selective peripheral vasopressors (without positive inotropic or chronotropic effects) could have deleterious effects on CO. Thus, it seems important to use a combined analysis of MAP and CO to estimate the afterload-related cardiac performance (ACP) The investigators recently proposed a cardiac afterload monitoring, in the descending thoracic aorta, based on a combined analysis of flow velocity signal recorded by trans-oesophageal Doppler and aortic pressure, the Velocity-Pressure Loop (VP Loop). VP Loop, and its derived indicators, especially Global AfterLoad Angle (GALA), could be useful during hemodynamic management for continuous cardiac afterload monitoring. However, in cardiology unit, cardiac afterload is usually measured at the ascending aorta behind the aortic valves.

The main objective of this study is to compare VP Loop parameters build in the ascending and descending thoracic aorta according to patient cardiovascular risk factors.

DETAILED DESCRIPTION:
Main objective In order to personalize patient approach and better care during surgery, the investigators recently proposed a cardiac afterload monitoring, in the descending thoracic aorta, based on a combined analysis of flow velocity signal recorded by trans-oesophageal Doppler and aortic pressure, the Velocity-Pressure Loop (VP Loop). Cardiac afterload is usually measured at the ascending aorta behind the aortic valves. The main objective of this study is then to compare VP Loop parameters build in the ascending and descending thoracic aorta according to patient cardiovascular risk factors.

Cardiac afterload is measured under general anesthesia in the ascending and descending aorta, using recognized arterial indices describing it and parameters derived from the VP loop.

Cardiac afterload can be schematically defined by the combination of three components: peripheral vascular resistance (PVR), total arterial compliance (Ctot) and aortic wave reflections (WR). WR could be assessed by pulse wave pressure analysis with the augmentation index (Aix) or after pulse wave pressure separation into a forward and backward wave with the wave reflection index (WRi) or the wave reflection area (WRa).

Aortic pressure measurements As required by the standard of care of the interventional neuroradiology procedure, the neuroradiologist also cannulated the femoral artery. At the end of the procedure, during catheter withdrawal, pressure waveforms are recorded at two predefined aortic locations: in the ascending aorta and in the descending thoracic aorta just in front of the esophageal Doppler probe.

Aortic velocity recording VP Loop in ascending aorta and aortic velocity are measured in the flushing chamber of the left ventricle from the apical five-chamber view by trans-thoracic echocardiography (TTE) (Philips, EPIQ 7). Descending aortic velocity is measured with a transesophageal Doppler CardioQ-ODM+ (Deltex Medical, Chichester, UK) in order to construct the VP Loop in descending thoracic aorta.

VP Loop construction Digitalization of pressure and velocity signals are performed with the IntelliVue MP60 monitor (Philips, Eindhoven, The Netherlands) at a sampling frequency of 125 Hz and saved using ixTrend software (ixellence, Wildau, Germany) on a computer.

Briefly, the velocity coordinates is plotted on the x axis and the pressure coordinates on the y axis. The investigators characterise the VP Loop by 4 points (A, B, C, D), allowing us to identify 3 angles: Alpha, Beta and GALA.

The goal of this study is to evaluate in patients cardiac after-load obtained by VP loop and to compare VP Loop parameters build in the ascending and descending thoracic aorta according to patient cardiovascular risk factors.

Experimental design This is a single-center, interventional, category II prospective study (minimal risks and constraints) Population concerned Patients will be included if their perioperative risk required a continuous monitoring of MAP and CO. The study involves major patients under general anaesthesia in interventional neuroradiology.

Research Proceedings For all patients, data from trans-oesophageal Doppler, trans-thoracic echocardiography (TTE) and hemodynamic data are collected at the end of the procedure. During catheter withdrawal, pressure waveforms are recorded at two predefined aortic locations: in the ascending aorta and in the descending thoracic aorta just in front of the esophageal Doppler probe. All data from monitoring are connected to the main monitor.

Individual benefit:

There is no benefit for the patient

Collective benefit:

Targeting mean arterial pressure (MAP) with boluses of selective peripheral vasopressors (without positive inotropic or chronotropic effects) could have deleterious effects on cardiac output. Thus, it seems important to use a combined analysis of MAP and CO with low invasive methods to estimate the Afterload-related cardiac performance (ACP) in surgical patients considered with "high cardiovascular risk".

Risks and minimal constraints added by the research No added risk. Patients are included if their perioperative risk required a continuous monitoring of MAP and CO. The standard of care for the interventional neuroradiology procedure needs a catheterization of the femoral artery using the Seldinger technique and insertion of a catheter. All the other ones measures are obtained non-invasively.

Patients are assigned to one of two groups according to their risk of increased arterial stiffness as reported in cardiological publications. The criteria used by investigators are as follows: age > 50 years old as a major criterion 20 and cardio-vascular risk factors (history of congestive heart failure, history of cardiovascular event, current smoking, diabetes mellitus, dyslipidemia, and arterial hypertension) as minor criteria. Patients were classified into the high risk group (Hi-risk) if they had at least one major criterion or two minor criteria or into the low risk group (Lo-risk) if they presented with no or one minor criterion.

During their interventional neuroradiology procedure, all patients' routine monitoring will consist of electrocardiogram, pulsated oxygen saturation, end-tidal CO2, respiratory rate, tidal volume and monitoring of neuromuscular function.

For all patients whatever the comorbidities, anesthesia induction will be performed using a target-controlled infusion (Orchestra® Base Primea - Fresenius Kabi France).

According to our standard of care, intra-operative episodes of hypotension (mean arterial pressure (MAP) < 65 mmHg or < 80% baseline) are treated by Norepinephrine bolus of 10 µg.

For all patients, data from trans-oesophageal Doppler, trans-thoracic echocardiography (TTE) and hemodynamic data are collected at the end of the procedure. During catheter withdrawal, pressure waveforms are recorded at two predefined aortic locations: in the ascending aorta and in the descending thoracic aorta just in front of the esophageal Doppler probe.

Number of selected subjects Selection of patients up to 55 analysable patients Number of Centre : 1 Research Agenda inclusion period: 12 months duration of participation (treatment + follow-up): duration of the interventional neuroradiology procedure: 1 day total duration: 12 months Number of planned inclusions by centre and month : 5 Number of subjects required : 55 Statistics

Continuous variables will be expressed as mean ± SD and qualitative variables are expressed as n (%). For comparison between LR and HR, investigators used the t-test or chi-squared test for continuous or categorical variables. The comparison of hemodynamic parameters between ascending and descending aorta is performed by a paired t-test. A Pearson correlation is used to study the relationship between different hemodynamic indices. Receiver operating characteristic curves (ROC) and Area under the curves (AUC) will be performed to calculate the performance of each cardiac afterload index to discriminate LR and HR patients. P-value less than 5% is considered significant.

The sample size calculation is based on the following assumptions: incidence of Hi-risk patients of 50%, as previously reported, incidence of increase of intrinsic arterial stiffness (after-load). In low risk patients a difference in arterial stiffness between low- and high-risk patients at 30%, power at 80% and type I error at 5%. Accordingly, the calculated sample size is 55 patients for the entire population.

ELIGIBILITY:
Inclusion Criteria:

* • Patients > 18 years scheduled an elective interventional neuroradiology procedure under general anesthesia requiring a continuous monitoring of mean arterial pressure and cardiac output.

  * oral agreement obtained from each patient before anesthesia

Exclusion Criteria:

* • age <18 years

  * an emergency procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with scheduled an elective interventional neuroradiology procedure under general anesthesia requiring a continuous monitoring of mean arterial pressure and cardiac output.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
Measure of aortic pressure in the ascending aorta and in the descending thoracic aorta in mmHg (PAo) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)]
  For all patients, aortic pressure will be collected at the end of the procedure during catheter withdrawal
Aortic velocity in the ascending aorta in cm/s (VAasc.) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, aortic ascending velocity will be collected at the end of the procedure during catheter withdrawal
Aortic velocity in the descending aorta in cm/s (VAdes.) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)]
  For all patients, aortic descending velocity will be collected at the end of the procedure during catheter withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Principal Investigator — HLariboisière